CLINICAL TRIAL: NCT06739187
Title: Virtual Reality Training for Cognitive Impairment in Adults Treated With Hemodialysis: A Feasibility Randomized Controlled Trial
Brief Title: Virtual Reality for Cognitive Impairment in Hemodialysis
Acronym: VIRTUAL
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Collaborators: University of Sydney (Other); University of Bari Aldo Moro (Other); University of Otago (Other)
Responsible Party: Principal Investigator, Davide Viggiano, Prof, University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRIN20225JEHW8; PRIN20225JEHW8 (Other Grant/Funding Number: PRIN 2022)
Record Dates: First submitted 2024-12-08; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Hemodialysis
Keywords: hemodialysis; virtual reality; RCT; kidney failure
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality (Active Comparator): Participants will use the virtual reality during the standard dialysis session for 30 minutes, three times a week for 12 weeks.
  Interventions: Device: Virtual reality platform on head mounted display
- Standard care (No Intervention): Participants will perform the standard dialysis session three times a week for 12 weeks without virtual reality training sessions.

INTERVENTIONS:
Device: Virtual reality platform on head mounted display — Enhance Virtual Reality platform on a Meta Quest head mounted display
  Arms: Virtual reality

SUMMARY:
The goal of this randomized feasibility clinical trial is to identify participant recruitment and retention, acceptability, and adherence to virtual reality training in people undergoing hemodialysis. The main question it aims to answer is if virtual reality could be a feasible and acceptable intervention in this setting.

The investigators will compare participants on virtual reality training during the standard dialysis session with those treated with standard dialysis session alone to see if a cognitive training using immersive virtual reality in people on hemodialysis is feasible and acceptable.

Participants randomised in the intervention group will use virtual reality during the standard dialysis session for 30 minutes, three times a week for 12 weeks. The virtual reality intervention will consist of computerized cognitive training of 4 games. Each exercise delivered to the participant will specifically provide training in a specific cognitive category (memory, cognitive flexibility, processing, attention, and memory). Participants randomised in the control group will perform the standard hemodialysis session three times a week for 12 weeks, without using virtual reality.

DETAILED DESCRIPTION:
The trial is a multicenter, parallel group, feasibility randomized controlled trial.

The trial population will include adult participants, who have the physical and cognitive capacity to be trained using immersive virtual reality and who have kidney failure on hemodialysis.

Participants will be allocated in the intervention (virtual reality session) or standard of care without the intervention. Participants will be allocated to intervention or standard care by randomization 1:1.

The virtual reality intervention will consist of computerized cognitive training of a subset of 4 short, gamified exercises. The intervention will be accessed through the Enhance VR platform on a Meta Quest 3S head mounted display, Snapdragon XR2 Gen2, processor, 8 Gb RAM, 128 Gb internal memory, resolution per eye in pixels: 1832 x 1920 with a refresh rate of 90-120 Hz and motion controllers. The clinician responsible for the intervention will be in the room with the participant, providing support for the intervention and any technical issues.

The chosen trial duration of 12 weeks is designed to provide exposure to a meaningful dose of cognitive training (three times a week) aligned to previous similar studies and to maximize participant tolerability to immersive virtual reality training.

The endpoints described in this protocol align with the recommendations of the CONSORT 2010 statement: extension to randomized pilot and feasibility studies. The endpoints are specifically chosen to relate to feasibility. The outcomes also include the primary and secondary outcomes for the future definitive randomized controlled trial to assess response, feasibility of measurement, and completeness.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants aged 18 years or older and less than or equal to 75 years of age
* Receiving haemodialysis treatment for kidney failure for at least 90 days (permanent reduction in kidney function below an estimated glomerular filtration rate of 15 mL/minute per 1.73 m2)
* Able to provide written and informed consent
* Able to use the immersive virtual reality headset and follow instructions with sufficient motor, visual and auditory function to interact with the intervention
* Able to speak and understand Italian language

Exclusion Criteria:

* Severe cognitive impairment or psychiatric diseases leading to inability to follow instructions and use the virtual reality headset
* Significant nystagmus and/or vertigo leading to inability to tolerate the virtual reality headset
* Insufficient motor function to use the virtual reality system
* Hearing or visual disability
* Advanced or uncompensated chronic diseases unrelated to kidney failure (e.g. advanced cancer, heart failure, lung diseases with poor oxygen saturation)
* Other neurological diseases (ictus, Alzheimer's or other forms of dementia)
* Persistent pain or itch or who using opioids that may interfere with the tests or any other condition that the clinician may judge as influencing the results

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Accept the invitation to participate | 4, 12 weeks
  Proportion of screened patients who participate in one or more sessions of allocated virtual reality training.
Appropriateness of eligibility criteria | 12 weeks
  Recruitment rate during 12 weeks of recruitment phase.
Retention | 12 weeks
  Proportion of randomized participants who complete the intervention and complete follow-up at 12 weeks.
Acceptability | 12 weeks
  Proportion of randomized participants who complete >80% of the treatments during 12 weeks follow-up.
Proportion of adverse events | 12 weeks
  Proportion of randomized participants who have adverse event reporting completed at 12 weeks.
Quality of life | 0, 4, 12, 24 weeks
  Proportion of randomized participants who complete the outcome measurements using the Kidney Disease Quality of Life Short Form 36 (KDQOL-36). The KDQOL-36 has five scales, including two generic health related quality of life scales from the SF-12 version 1 (12 items total) and three kidney-specific scales (24 items total). Each of the KDQOL-36 kidney-targeted scales are scored by transforming all items linearly to a 0-100 possible range and averaging the items in the scale. On the KDQOL-36, higher scores indicate better health realated quality of life.

SECONDARY OUTCOMES:
Depression | 0, 4, 12, 24 weeks
  Proportion of randomized participants who complete the outcome measurements using the Hospital Anxiety and Depression Scale (HADS). The HADS consists of 14 items, divided in two seven-item subscales. The total score for each subscale ranges from 0 to 21. In general a score ≤7 corresponds to "no depression or anxiety," a score of 8-10 is a minor depression/anxiety, a score of 11-15 a moderate depression/anxiety and a score ≥16 is defined as severe depression/anxiety.
Anxiety | 0, 4, 12, 24 weeks
  Proportion of randomized participants who complete the outcome measurements using the Hospital Anxiety and Depression Scale (HADS). The HADS consists of 14 items, divided in two seven-item subscales. The total score for each subscale ranges from 0 to 21. In general a score ≤7 corresponds to "no depression or anxiety," a score of 8-10 is a minor depression/anxiety, a score of 11-15 a moderate depression/anxiety and a score ≥16 is defined as severe depression/anxiety.
Quality of life | 0, 4, 12, 24 weeks
  Proportion of randomized participants who complete the outcome measurements using the 5-level EQ-5D version (EQ-5D-5L). In the EQ-5D-5L scores range from 0 to 100, where 100 is the best possible health related quality of life.
Fatigue | 0, 4, 12, 24 weeks
  Proportion of randomized participants who complete the outcome measurements using the Kidney Disease Quality of Life Short Form 36 (KDQOL-36). The KDQOL-36 has five scales, including two generic health related quality of life scales from the SF-12 version 1 (12 items total) and three kidney-specific scales (24 items total). Each of the KDQOL-36 kidney-targeted scales are scored by transforming all items linearly to a 0-100 possible range and averaging the items in the scale. On the KDQOL-36, higher scores indicate better outcome.
Health utility | 0 and 12 weeks
  Proportion of randomized participants who complete an authors' designed questionnaire
All-cause death | 12 weeks
  All-cause death reported during the study
Cardiovascular events | 12 weeks
  All cardiovascular events (myocardial infarction, stroke, peripheral arterial event) reported during the study
Pulse | 0 and 12 weeks
  Pulse rate (bpm)
Systolic blood pressure | 0 and 12 weeks
  Systolic blood pressure (mmHg)
Diastolic blood pressure | 0 and 12 weeks
  Diastolic blood pressure (mmHg)
Functional near-infrared spectroscopy | 0 and 12 weeks
  Functional near-infrared spectroscopy (fNIR)
Kt/V | 0 and 12 weeks
  Kt/V
Dialysis duration | 0 and 12 weeks
  Dialysis duration (min)
Type of dialysis | 0 and 12 weeks
  Type of dialysis
Hemoglobin | 0 and 12 weeks
  Hemoglobin (g/dL)
Glucose | 0 and 12 weeks
  Glucose (mg/dL)
Glycated hemoglobin | 0 and 12 weeks
  HbA1c (%)
Serum creatinine | 0 and 12 weeks
  Serum creatinine (mg/dL)
Serum albumin | 0 and 12 weeks
  Serum albumin (g/dL)

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - University of Bari, Bari, BA
  - Univerity Vanvitelli, Naples

IPD SHARING:
Plan to Share IPD: No
Data will be available after request to the principal investigator.